CLINICAL TRIAL: NCT05360069
Title: Linear Stapler Versus Circular Stapler in Esophagojejunostomy for Patients With Gastric Cancer Underwent Laparoscopic Total Gastrectomy
Brief Title: Linear Stapler Versus Circular Stapler in Esophagojejunostomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchong Central Hospital (Other Government)
Responsible Party: Principal Investigator, Yunhong Tian, Professor, Nanchong Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202101
Record Dates: First submitted 2022-03-11; First posted 2022-05-04 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Complications; Operative Time; Hospital Costs
Keywords: laparoscopy; total gastrectomy; esophagojejunostomy; linear stapler; circular stapler
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Linear stapler group (Experimental): Linear stapler is adopted in esophagojejunostomy.
  Interventions: Device: Linear stapler
- Circular stapler group (Active Comparator): Circular stapler is adopted in esophagojejunostomy.
  Interventions: Device: Circular stapler

INTERVENTIONS:
Device: Linear stapler — Linear stapler is adopted in esophagojejunostomy
  Arms: Linear stapler group
Device: Circular stapler — Circular stapler is adopted in esophagojejunostomy
  Arms: Circular stapler group

SUMMARY:
With the development of stapler devices, various methods of esophagojejunostomy after laparoscopic total gastrectomy were evoluated. Which stapler is more advantageous has not been determined. At present, the most commonly used is linear stapler or Circular stapler in esophagojejunostomy. However, there is still a lack of reliable evidence for the selection of the two staplers. The purpose of this study is to explore the advantages of linear staper versus circular stapler in esophagojejunostomy for patients with gastric cancer who underwent total gastrectomy.

DETAILED DESCRIPTION:
With the development of stapler devices, various methods of esophagojejunostomy after laparoscopic total gastrectomy were evoluated. Which stapler is more advantageous has not been determined. At present, the most commonly used is linear stapler or Circular stapler in esophagojejunostomy. However, there is still a lack of reliable evidence for the selection of the two staplers. The purpose of this study is to explore the advantages of linear staper versus circular stapler in esophagojejunostomy for patients with Siewert classification type II and III gastric cancer who underwent total gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the stomach, T1-T4 stages.
2. Eastern Cooperative Oncology Group performance status of 0 or 1.
3. Adequate organ function.

Exclusion Criteria:

1. Patients had distant metastasis.
2. oesophageal invasion of more than 3 cm.
3. Borrmann type 4 or large (more than 8 cm) type 3 carcinoma.
4. Previous chemotherapy or radiation therapy for any other malignancies.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical complication | 6 months
  All surgical complication after laparoscopic total gastrectomy

SECONDARY OUTCOMES:
Operation duration | 1 day
  operation time

OTHER OUTCOMES:
hospitalization cost | 2 months
  the cost in hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Yunhong Tian, Nanchong, Sichuan, China